CLINICAL TRIAL: NCT01145911
Title: The Study of Ocular Hemodynamics With Glaucoma Progression
Acronym: IGPS
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Other Study IDs: IGPS
Record Dates: First submitted 2010-06-15; First posted 2010-06-17 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Glaucoma
Keywords: Glaucoma; Blood Flow; Progression
MeSH Terms: conditions — Glaucoma; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Glaucoma patients: Glaucoma patients

SUMMARY:
To determine the relationships between ocular hemodynamics and glaucomatous optic neuropathy progression.

DETAILED DESCRIPTION:
1. To determine whether baseline ocular blood flow values are predictive of glaucomatous progression as determined by visual field analysis.
2. To determine how changes in ocular blood flow are related to visual field progression.
3. To determine how changes in ocular blood flow are related to changes in optic nerve structure and topographic change over time.

ELIGIBILITY:
Inclusion Criteria:

Patients will meet all of the following inclusion criteria to enter the study:

1. Age: 30 years or older.
2. Diagnosis: confirmed open-angle glaucoma in at least one eye:

   1. glaucomatous visual field loss on Humphrey 24-2 or 10-2 perimetry
   2. glaucomatous optic disc cupping
   3. agreement between two baseline exams for reliability
3. Best corrected visual acuity at least 20/60 in at least one eye.
4. Prior Humphrey visual fields demonstrate acceptable reliability standards (see below).

Exclusion Criteria:

1. Extensive Humphrey visual field damage consisting of either a mean deviation (MD) < -15 decibels or a clinically determined threat to fixation in both hemifields.
2. Evidence of exfoliation or pigment dispersion.
3. History of acute angle-closure or a narrow, occludable anterior chamber angle by gonioscopy.
4. History of chronic or recurrent inflammatory eye diseases (e.g., scleritis, uveitis).
5. History or signs of intraocular trauma.
6. Severe or potentially progressive retinal disease such as retinal degeneration, diabetic retinopathy, and retinal detachment.
7. Any abnormality preventing reliable applanation tonometry.
8. Current use of any ophthalmic or systemic steroid which may interfere with this investigation.
9. Cataract surgery within the past year.
10. Resting pulse < 50 beats per minute.
11. Severe, unstable or uncontrolled cardiovascular, renal, or pulmonary disease.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Glaucoma patients
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2008-01; Primary Completion 2014-07-03 (Actual); Study Completion 2014-07-03 (Actual)

PRIMARY OUTCOMES:
Ocular Blood Flow | various
  per visit

CONTACTS AND LOCATIONS:
Overall Officials: Alon Harris, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University School of Medicine, Department of Ophthalmology, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Verticchio Vercellin AC, Harris A, Oddone F, Siesky B, Eckert G, Belamkar A, Antman G, Segev F. Ocular blood flow biomarkers may predict long-term glaucoma progression. Br J Ophthalmol. 2024 Jun 20;108(7):946-950. doi: 10.1136/bjo-2022-322644. PMID 37852742